CLINICAL TRIAL: NCT03706352
Title: Postoperative Pain: Is Tunneling Effective in Preventing Failure of Epidural Analgesia? A Randomized Trial
Brief Title: Is Tunneling Effective in Preventing Failure of Epidural Analgesia? A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Hussein Abu Khudair, chairman department of anesthesiology and pain management, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13KHCC64
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Epidural Catheter; Post Operative Pain
Keywords: Cancer patients, Epidural analgesia, Postoperative pain, tunneling
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tunneling group (Experimental): Epidural Catheter Insertion and fixation by subcutaneous tunneling procedure.
  Interventions: Procedure: tunneling epidural catheter
- taping group (Active Comparator): Epidural Catheter Insertion and fixation by use of adhesive tape without tunneling.
  Interventions: Procedure: tunneling epidural catheter

INTERVENTIONS:
Procedure: tunneling epidural catheter — The epidural needle was used to horizontally tunnel the catheter for a length of five centimeters on either side of the insertion point.

SUMMARY:
This is a prospective randomized single blinded study in patients planned to undergo general anesthesia and epidural catheter insertion for pain control after abdominal, thoracic and orthopedic surgery.

Patients meeting participation criteria will be selected and enrolled sequentially.

The study recruitment will be carried out over one year with follow-up for each patient until either the catheter is dislodged or once decided that the patient is to be discontinued from the epidural pain control.

DETAILED DESCRIPTION:
Study Population and Sample Size The study aims to enroll 200 adult patients planned to undergo general anesthesia and epidural catheter insertion. The study sample will be selected to fulfill the selection criteria.

Patients will be selected if they meet the following participation criteria:

Planned Procedures and Assessments Follow -up on dislodgments, adverse events, pain and pain relief assessment, standard practice Study Site All study conduction from start to end including procedures and assessments, data acquisition and analysis and final study conclusion report and any publications will be at King Hussein Cancer Center (KHCC).

Ethical Considerations The study will be submitted to the KHCC IRB for review. The study will not start before IRB approval is obtained.

All patients who provide consent to participation in the study will be randomized and enrolled.

Statistical Plan Descriptive statistics will be used to present the two groups baseline characteristics. Comparison between groups will be carried out using Chi-square test or t-test or Wilcox on rank test as appropriate. Comparison between groups while adjusting for other variables will be carried out using logistic regression. Odds ratios along with their 95% confidence intervals will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult, between 18-80 years old with normal mentation.

  * Patient has consented to general anesthesia and epidural catheter insertion for pain control after abdominal, thoracic and orthopedic surgery
  * Patient is able to understand and provide informed consent to participate in the study.

Exclusion Criteria:

Patient is prone to coagulopathy.

* Patient has infection at injection site.
* Any Patient seen immediately before surgery-

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Difference in Rate of dislodgment between the two groups | 5 days
  Descriptive statistics will be used to present the two groups baseline characteristics. Comparison between groups will be carried out using Chi-square test or t-test or Wilcox on rank test as appropriate. Comparison between groups while adjusting for other variables will be carried out using logistic regression. Odds ratios along with their 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
standard numerical pain score (NPS) | 5 days
  use numerical pain score from zero no pain and 10 worst immaginable pain
Rate of adverse events | 5 days
  infection, pain bleeding nerve damage, headache

IPD SHARING:
Plan to Share IPD: No